CLINICAL TRIAL: NCT02864251
Title: Open-Label, Randomized Trial of Nivolumab (BMS-936558) Plus Pemetrexed/Platinum or Nivolumab Plus Ipilimumab (BMS-734016) vs Pemetrexed Plus Platinum in Stage IV or Recurrent Non-Small Cell Lung Cancer (NSCLC) Subjects With Epidermal Growth Factor Receptor (EGFR) Mutation Who Failed 1L or 2L EGFR Tyrosine Kinase Inhibitor Therapy
Brief Title: A Study of Nivolumab + Chemotherapy or Nivolumab + Ipilimumab Versus Chemotherapy in Non-Small Cell Lung Cancer (NSCLC) Participants With Epidermal Growth Factor Receptor (EGFR) Mutation Who Failed 1L or 2L EGFR Tyrosine Kinase Inhibitor (TKI) Therapy
Acronym: CheckMate722
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-722; 2017-002672-38 (EudraCT Number)
Record Dates: First submitted 2016-08-09; First posted 2016-08-11 (Estimated); Results first posted 2023-02-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nivolumab+Platinum doublet chemotherapy (Experimental)
  Interventions: Biological: Nivolumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Nivolumab + Ipilimumab (Experimental): Enrollment is closed for this arm
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Platinum doublet chemotherapy (Active Comparator)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Nivolumab + Ipilimumab; Nivolumab+Platinum doublet chemotherapy
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
  Arms: Nivolumab + Ipilimumab
Drug: Pemetrexed — Specified dose on specified days
  Arms: Nivolumab+Platinum doublet chemotherapy; Platinum doublet chemotherapy
Drug: Cisplatin — Specified dose on specified days
  Arms: Nivolumab+Platinum doublet chemotherapy; Platinum doublet chemotherapy
Drug: Carboplatin — Specified dose on specified days
  Arms: Nivolumab+Platinum doublet chemotherapy; Platinum doublet chemotherapy

SUMMARY:
The main purpose of this study is to determine whether nivolumab + chemotherapy is effective as compared to chemotherapy in the treatment of patients with EGFR mutation, NSCLC who failed first line (1L) or second-line (2L) EGFR TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed stage IV or recurrent EGFR mutated NSCLC with disease progression on one or two prior lines of treatment with EGFR TKIs (allowed TKIs must be approved by the local health authority, including but not limited to erlotinib, gefitinib, afatinib, dacomitinib and osimertinib). In osimertinib treated subjects, T790 testing is not required.
* No evidence of exon 20 T790M mutation obtained at progression on prior first- or second-generation EGFR TKI therapy. For participants who were treated with osimertinib, T790M testing is not required.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Available tumor sample for Programmed death-ligand 1 (PD-L1) immunohistochemical (IHC).
* Participants are eligible if central nervous system (CNS) metastases are considered to be adequately controlled/treated before or during the screening period and participants are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to randomization. In addition, participants must be either off corticosteroids, or on a stable or decreasing dose of ≤10 mg daily prednisone (or equivalent) for at least 2 weeks prior to randomization). Participants with asymptomatic CNS metastasis are eligible.
* Eastern Cooperative Group (ECOG) Performance Status 0-1
* Life expectancy is at least 3 months

Exclusion Criteria:

* Known EGFR mutation, T790M positive who failed 1L first- or second-generation TKI should receive osimertinib first as the standard of care (SOC). These participants are only eligible if they fail osimertinib as 2L.
* who have progressed within 3 months of the first dose of 1L or 2L EGFR TKI.
* Carcinomatous meningitis
* Active, known or suspected autoimmune disease are excluded
* ALK translocation
* Known SCLC transformation
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (102):
- United States (18):
  - Pacific Shores Medical Group, Long Beach, California
  - Local Institution - 0029, Los Angeles, California
  - Local Institution - 0033, Los Angeles, California
  - Local Institution - 0061, Orange, California
  - Torrance Memorial Physican Network, Redondo Beach, California
  - Local Institution - 0003, New Haven, Connecticut
  - Local Institution - 0004, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Local Institution - 0002, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 0064, New York, New York
  - Duke University Medical Center, Butner, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Health Physicians Group, Arlington, Texas
  - Baylor Scott and White Research Institute, Temple, Texas
  - Local Institution - 0063, Tyler, Texas
  - Local Institution - 0001, Salt Lake City, Utah
- Canada (2):
  - Local Institution - 0166, Edmonton, Alberta
  - Local Institution - 0168, Montreal, Quebec
- China (13):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Zhengzhou, Henan
  - Local Institution, Hong Kong, HONG KONG
  - Local Institution - 0043, Changsha, Hunan
  - Local Institution, Changchun, Jilin
  - Local Institution, Xi'an, Shan3xi
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution - 0016, Hangzhou, Zhejiang
  - Local Institution - 0017, Hangzhou, Zhejiang
  - Local Institution, Hangzhou, Zhejiang
- France (4):
  - Local Institution, Marseille
  - Local Institution - 0156, Paris
  - Local Institution, Rennes
  - Local Institution, Toulouse
- Hong Kong (3):
  - Local Institution - 0027, Hong Kong
  - Local Institution - 0024, Hong Kong
  - Local Institution, Shatin
- Japan (34):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Hirosaki-shi, Aomori
  - Local Institution, Matsuyama, Ehime
  - Local Institution, Iizuka, Fukuoka
  - Local Institution - 0059, Kurume, Fukuoka
  - Local Institution, Fukushima, Fukushima
  - Local Institution, Kōriyama, Fukushima
  - Local Institution, Fukuyama, Hiroshima
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution - 0070, Sapporo, Hokkaido
  - Local Institution, Himeji-shi, Hyōgo
  - Local Institution - 0097, Itami, Hyōgo
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Bunkyō City, Kanagawa
  - Local Institution - 0081, Yokohama, Kanagawa
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Natori-shi, Miyagi
  - Local Institution - 0077, Sendai, Miyagi
  - Local Institution, Hirakata-shi, Osaka
  - Local Institution, Kishiwada Shi, Osaka
  - Local Institution, Sakai, Osaka
  - Local Institution - 0058, Sayama, Osaka
  - Local Institution - 0076, Hidaka, Saitama
  - Local Institution, Kitaadachi-gun, Saitama
  - Local Institution - 0069, Chūō, Tokyo
  - Local Institution - 0078, Koto-ku, Tokyo
  - Local Institution, Ube Shi, Yamaguchi
  - Local Institution, Chiba
  - Local Institution, Fukuoka
  - Local Institution, Niigata
  - Local Institution - 0079, Tokyo
  - Local Institution, Toyama
  - Local Institution, Wakayama
- Singapore (2):
  - Local Institution - 0042, Singapore
  - Local Institution - 0041, Singapore
- South Korea (8):
  - Local Institution - 0038, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0037, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0035, Seoul, Seoul Teugbyeolsi
  - Local Institution, Cheogju-si
  - Local Institution, Gyeonggi-do
  - Local Institution - 0036, Gyeonggi-do
  - Local Institution, Inchoen
  - Local Institution, Seoul
- Spain (6):
  - Local Institution - 0158, Barcelona
  - Local Institution, L'Hospitalet de Llobregat
  - Local Institution, Madrid
  - Local Institution, Majadahonda
  - Local Institution, Málaga
  - Local Institution, Zaragoza
- Taiwan (12):
  - Local Institution - 0021, Tainan, TNN
  - Local Institution - 0045, Chiayi City
  - Local Institution, Kaohsiung City
  - Local Institution - 0019, Kaohsiung City
  - Local Institution - 0018, Taichung
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
  - Local Institution - 0066, Taipei
  - Local Institution - 0108, Taipei
  - Local Institution - 0023, Taipei
  - Local Institution, Taoyuan District

REFERENCES:
- [Derived] Mok T, Nakagawa K, Park K, Ohe Y, Girard N, Kim HR, Wu YL, Gainor J, Lee SH, Chiu CH, Kim SW, Yang CT, Wu CL, Wu L, Lin MC, Samol J, Ichikado K, Wang M, Zhang X, Sylvester J, Li S, Forslund A, Yang JC. Nivolumab Plus Chemotherapy in Epidermal Growth Factor Receptor-Mutated Metastatic Non-Small-Cell Lung Cancer After Disease Progression on Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors: Final Results of CheckMate 722. J Clin Oncol. 2024 Apr 10;42(11):1252-1264. doi: 10.1200/JCO.23.01017. Epub 2024 Jan 22. PMID 38252907
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arm B: Nivolumab plus Ipilimumab was exploratory and closed prior to primary completion.
Groups:
- Arm A: Nivolumab Plus Platinum-doublet Chemotherapy: Nivolumab was administered IV every 3 weeks with platinum-doublet chemotherapy (investigator's choice of cisplatin or carboplatin) IV for a maximum of 4 cycles.
  Treatment administered was either Nivolumab 360 mg IV, followed by pemetrexed (500 mg/m2) with cisplatin (75 mg/m2) administered on Day 1 of each cycle OR Nivolumab 360 mg IV, followed by pemetrexed (500 mg/m2) with carboplatin (AUC 5 or 6) administered on Day 1 of each cycle.
  Following completion of the fourth cycle of nivolumab/chemotherapy, all participants who did not experience disease progression should have continued nivolumab 360 mg IV and pemetrexed (500 mg/m2) every 3 weeks until the progression of disease, discontinuation due to toxicity, withdrawal of consent, or study closure, whichever comes first. Nivolumab should only be administered for a maximum of 24 months (96 weeks) from the first study treatment.
- Arm B: Nivolumab Plus Ipilimumab: Nivolumab 3 mg/kg IV was administered every 2 weeks and ipilimumab 1 mg/kg IV was administered every 6 weeks until the progression of disease, discontinuation due to toxicity, withdrawal of consent, a maximum of 24 months (96 weeks) from the first study treatment, or study closure.
- Arm C: Platinum Doublet Chemotherapy: Platinum-doublet chemotherapy (investigator's choice of cisplatin or carboplatin) was administered IV in 3-week cycles for up to a maximum of 4 cycles.
  Participants received either Pemetrexed (500 mg/m2) with cisplatin (75 mg/m2) administered on Day 1 of each cycle OR Pemetrexed (500 mg/m2) with carboplatin (AUC 5 or 6) administered on Day 1 of each cycle.
  Platinum-doublet chemotherapy continued until disease progression, unacceptable toxicity, or completion of the 4 cycles, whichever came first.
  Participants who had stable disease or response after 4 cycles of pemetrexed with cisplatin or carboplatin should have continued pemetrexed alone as maintenance therapy until disease progression, or unacceptable toxicity.
Period: Pre-Treatment
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy
Started (Started = Randomized) | 144 | 73 | 150
Completed (Completed = Started Treatment) | 141 | 71 | 143
Not Completed | 3 | 2 | 7
Not completed — Adverse Event Unrelated to Study drug | 1 | 0 | 0
Not completed — Withdrawal by Participant | 0 | 0 | 4
Not completed — Participant no Longer Meets Study Criteria | 2 | 1 | 2
Not completed — Other Reasons | 0 | 1 | 1
Period: Treatment
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy
Started (Started Treatment) | 141 | 71 | 143
Completed (Completed Treatment) | 3 | 5 | 0
Not Completed | 138 | 66 | 143
Not completed — Disease Progression | 109 | 52 | 101
Not completed — Study Drug Toxicity | 9 | 4 | 10
Not completed — Death | 0 | 2 | 3
Not completed — Adverse Event Unrelated to Study Drug | 1 | 1 | 6
Not completed — Participant Requested to Discontinue Study Treatment | 8 | 0 | 5
Not completed — Withdrawal by Participant | 8 | 5 | 13
Not completed — Maximum Clinical Benefit | 1 | 0 | 1
Not completed — Participant no Longer Meets Study Criteria | 0 | 1 | 0
Not completed — Other Reasons | 1 | 1 | 4
Not completed — Administrative Reason by Sponsor | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy | Total
Number analyzed (Participants) | 144 | 73 | 150 | 367
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (10.6) | 61.9 (10.6) | 60.7 (10.1) | 61.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 37 | 94 | 214
  Male | 61 | 36 | 56 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 59 | 39 | 73 | 171
  Unknown or Not Reported | 85 | 34 | 77 | 196
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 136 | 68 | 139 | 343
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 3 | 11 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Blinded Independent Centralized Review (BICR)
Description: PFS is defined as the time between the date of randomization and the date of first documented tumor progression, as determined by BICR (per RECIST v1.1 criteria), or death due to any cause, whichever occurs first.
  Participants who died without reported progression will be considered to have progressed on the date of their death. Subsequent therapy was accounted for by censoring at the last evaluable tumor assessment on or prior to the date of subsequent therapy.
  Progression is the appearance of one or more new lesions. RECIST - "response evaluation criteria in solid tumors" is a standard system to measure tumor response to treatment.
  Based on Kaplan-Meier estimates
Time Frame: From randomization to the date of first documented tumor progression or death (approximately 58 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy
Number analyzed (Participants) | 144 | 73 | 150
Months | 5.59 [4.47 to 6.80] | 1.54 [1.41 to 2.63] | 5.45 [4.40 to 5.65]
Statistical Analysis 1: Comparison: Arm A: Nivolumab Plus Platinum-doublet Chemotherapy vs Arm C: Platinum Doublet Chemotherapy; Test type: Superiority; p = 0.0528, Log Rank — Log-rank test stratified by PD-L1 expression (>= 1% vs <1%/indeterminate/not evaluable), brain metastases (presence vs absence), smoking history (current/former vs never smoker), and prior osimertinib use (yes vs no) from IRT; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.56 to 1.00] — Arm A over Arm C Stratified Cox proportional hazard model
Statistical Analysis 2: Comparison: Arm B: Nivolumab Plus Ipilimumab vs Arm C: Platinum Doublet Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 2.07, 95% CI 2-sided [1.43 to 2.99] — Arm B over Arm C Stratified Cox proportional hazard model

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time between the date of randomization and the date of death due to any cause. OS will be censored on the last date a participant was known to be alive.
  Median based on Kaplan-Meier Estimates
Time Frame: From randomization to the date of death due to any cause (up to approximately 67 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy
Number analyzed (Participants) | 144 | 73 | 150
Months | 19.35 [16.13 to 20.99] | 17.12 [13.67 to 23.59] | 15.90 [14.00 to 18.79]
Statistical Analysis 1: Comparison: Arm A: Nivolumab Plus Platinum-doublet Chemotherapy vs Arm C: Platinum Doublet Chemotherapy; Test type: Superiority; p = 0.2180, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.62 to 1.12] — Hazard Ratio (Arm A over Arm C) is based on a stratified Cox proportional hazard model
Statistical Analysis 2: Comparison: Arm B: Nivolumab Plus Ipilimumab vs Arm C: Platinum Doublet Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.75 to 1.52] — Hazard Ratio (Arm B over Arm C) is based on a stratified Cox proportional hazard model

3. Secondary Outcome: Objective Response Rate (ORR) by Blinded Independent Centralized Review (BICR)
Description: ORR is number of randomized participants who have confirmed best overall response (BOR) of complete response (CR) or partial response (PR) using RECIST v1.1 criteria by BICR assessment.
  BOR is the best response designation, between randomization and objectively documented progression per RECIST v1.1 criteria by BICR or the date of subsequent anti-cancer therapy, whichever occurs first.
  PR is at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as reference. CR is disappearance of all target lesions and a reduction in the short axis of pathological lymph nodes to <10 mm (whether target or non-target).
  Radiographic tumor response assessments from Week 7 (± 7 days), then every 6 weeks (± 7 days) until Week 49 and every 12 weeks (± 7 days) thereafter, until disease progression, treatment discontinued, or the start of subsequent anti-cancer therapy.
  CR+PR, confidence interval based on the Clopper and Pearson method.
Time Frame: From randomization to the date of objectively documented progression, date of death, or the date of subsequent therapy (up to approximately 67 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy
Number analyzed (Participants) | 144 | 73 | 150
Percent of Participants | 30.6 [23.2 to 38.8] | 13.7 [6.8 to 23.8] | 26.7 [19.8 to 34.5]
Statistical Analysis 1: Comparison: Arm A: Nivolumab Plus Platinum-doublet Chemotherapy vs Arm C: Platinum Doublet Chemotherapy; Test type: Superiority; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.75 to 2.16] — Strata adjusted odds ratio (Arm A over Arm C) using Mantel-Haenszel method

4. Secondary Outcome: Duration of Response (DOR) by Blinded Independent Centralized Review (BICR)
Description: DOR is the time between the date of first response (CR or PR) and the date of first documented disease progression as determined by Response Evaluation Criteria In Solid Tumors (RECIST 1.1) or death due to any cause (death occurring after re-treatment or randomization to new combination treatment was not included), whichever occurred first.
  PR is at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as reference. CR is disappearance of all target lesions and a reduction in the short axis of pathological lymph nodes to <10 mm (whether target or non-target).
  Radiographic tumor response assessments from Week 7 (± 7 days), then every 6 weeks (± 7 days) until Week 49 and every 12 weeks (± 7 days) thereafter, until disease progression, treatment discontinued, or the start of subsequent anti-cancer therapy.
  Participants who neither progress nor die were censored on the date of their last assessment.
  Median computed using Kaplan-Meier method
Time Frame: From randomization to the date of first documented disease progression or death due to any cause (approximately 67 months)
Population: Randomized participants with CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy
Number analyzed (Participants) | 44 | 10 | 40
Months | 6.67 [4.17 to 12.45] | 50.04 [2.86 to NA] — Insufficient number of participants with events | 5.55 [4.07 to 9.92]

5. Secondary Outcome: 9 Month Progression Free Survival Rates (PFSR) by Blinded Independent Centralized Review (BICR)
Description: The PFSR at 9 months is defined as the percent of treated participants remaining progression free and surviving at 9 months since the first dosing date. Progression is the appearance of one or more new lesions.
  Point estimates are derived from Kaplan-Meier analyses.
Time Frame: 9 months after first treatment dose
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy
Number analyzed (Participants) | 144 | 73 | 150
Percent of Participants | 25.9 [18.4 to 34.0] | 12.2 [5.5 to 21.7] | 19.8 [12.6 to 28.1]

6. Secondary Outcome: 12 Month Progression Free Survival Rates (PFSR) by Blinded Independent Centralized Review (BICR)
Description: The PFSR at 12 months is defined as the percent of treated participants remaining progression free and surviving at 12 months since the first dosing date. Progression is the appearance of one or more new lesions. Point estimates are derived from Kaplan-Meier analyses.
Time Frame: 12 Months after first treatment dose
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy
Number analyzed (Participants) | 144 | 73 | 150
Percent of Participants | 21.2 [14.3 to 29.1] | 12.2 [5.5 to 21.7] | 15.9 [9.3 to 24.0]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion (up to approximately 67 months.) SAEs and Other AEs was assessed from first dose to 100 days post the last dose of study therapy (up to approximately an average of 11 months and a maximum of 51 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study therapy or similar.
Arm/Group | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy | Arm B: Nivolumab Plus Ipilimumab | Arm C: Platinum Doublet Chemotherapy
All-Cause Mortality (participants affected / at risk) | 92/144 | 55/73 | 105/150
Serious Adverse Events (participants affected / at risk) | 77/141 | 46/71 | 55/143
Other Adverse Events (participants affected / at risk) | 136/141 | 62/71 | 140/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy (N=141) | Arm B: Nivolumab Plus Ipilimumab (N=71) | Arm C: Platinum Doublet Chemotherapy (N=143)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Immune-mediated myocarditis (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0
Thyroiditis subacute (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 1
Catheter site oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 2 | 1
Sudden death (General disorders) | 1 | 1 | 0
Swelling (General disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 2 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 1
Breast cellulitis (Infections and infestations) | 0 | 0 | 1
Carbuncle (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 10 | 4 | 7
Pneumonia aspiration (Infections and infestations) | 2 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatine increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Platelet count decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 | 20 | 22
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab Plus Platinum-doublet Chemotherapy (N=141) | Arm B: Nivolumab Plus Ipilimumab (N=71) | Arm C: Platinum Doublet Chemotherapy (N=143)
Anaemia (Blood and lymphatic system disorders) | 66 | 7 | 58
Neutropenia (Blood and lymphatic system disorders) | 22 | 3 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 1 | 6
Hyperthyroidism (Endocrine disorders) | 7 | 8 | 0
Hypothyroidism (Endocrine disorders) | 15 | 12 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 11
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 4
Constipation (Gastrointestinal disorders) | 52 | 21 | 57
Diarrhoea (Gastrointestinal disorders) | 18 | 17 | 17
Nausea (Gastrointestinal disorders) | 63 | 12 | 60
Stomatitis (Gastrointestinal disorders) | 12 | 4 | 10
Vomiting (Gastrointestinal disorders) | 35 | 7 | 21
Asthenia (General disorders) | 12 | 3 | 10
Face oedema (General disorders) | 8 | 0 | 9
Fatigue (General disorders) | 30 | 15 | 19
Malaise (General disorders) | 18 | 5 | 21
Non-cardiac chest pain (General disorders) | 10 | 7 | 8
Oedema peripheral (General disorders) | 26 | 8 | 18
Pyrexia (General disorders) | 29 | 14 | 17
Conjunctivitis (Infections and infestations) | 10 | 2 | 2
Nasopharyngitis (Infections and infestations) | 8 | 1 | 1
Paronychia (Infections and infestations) | 6 | 4 | 1
Pneumonia (Infections and infestations) | 7 | 5 | 7
Upper respiratory tract infection (Infections and infestations) | 9 | 6 | 9
Urinary tract infection (Infections and infestations) | 5 | 4 | 3
Alanine aminotransferase increased (Investigations) | 35 | 12 | 26
Amylase increased (Investigations) | 13 | 3 | 9
Aspartate aminotransferase increased (Investigations) | 35 | 11 | 27
Blood creatinine increased (Investigations) | 19 | 1 | 15
Neutrophil count decreased (Investigations) | 42 | 4 | 45
Platelet count decreased (Investigations) | 19 | 6 | 28
Weight decreased (Investigations) | 9 | 7 | 6
White blood cell count decreased (Investigations) | 38 | 3 | 35
Decreased appetite (Metabolism and nutrition disorders) | 42 | 16 | 52
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 | 2 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 6 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 9 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 5 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 5 | 9
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7 | 3
Dizziness (Nervous system disorders) | 15 | 7 | 14
Dysgeusia (Nervous system disorders) | 9 | 1 | 10
Headache (Nervous system disorders) | 22 | 5 | 19
Anxiety (Psychiatric disorders) | 6 | 4 | 3
Insomnia (Psychiatric disorders) | 17 | 6 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 16 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 14 | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 9
Hiccups (Respiratory, thoracic and mediastinal disorders) | 12 | 2 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 4 | 8
Eczema (Skin and subcutaneous tissue disorders) | 2 | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 18 | 8
Rash (Skin and subcutaneous tissue disorders) | 2 | 9 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 2 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 12 | 9 | 1
Hypertension (Vascular disorders) | 9 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02864251/Prot_SAP_000.pdf